CLINICAL TRIAL: NCT03711253
Title: Empiric Treatment for Suspected Acute HIV Infection in the Emergency Department
Brief Title: Empiric Treatment for Acute HIV in the ED
Acronym: EMTreatED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael Dube, Professor of Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-18-01821
Record Dates: First submitted 2018-07-26; First posted 2018-10-18 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Acute HIV Infection
Keywords: acute hiv infection; emergency department; antiretroviral therapy
MeSH Terms: conditions — Emergencies | interventions — bictegravir; Emtricitabine; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biktarvy (Other): All participants get Biktarvy Bictegravir 50mg+Tenofovir AF 25 mg+emtricitabine 200 mg in this single arm study
  Interventions: Drug: Bictegravir 50mg+Tenofovir AF 25 mg+emtricitabine 200 mg

INTERVENTIONS:
Drug: Bictegravir 50mg+Tenofovir AF 25 mg+emtricitabine 200 mg — antiretroviral therapy
  Other Names: Biktarvy

SUMMARY:
An acceptance and feasibility study for immediate ART initiation and storage of laboratory specimens for individuals with suspected acute HIV infection who are diagnosed in one of the 7 participating emergency rooms

DETAILED DESCRIPTION:
Individuals with suspected acute HIV infection willing to start immediate ART treatment will be given the ART regimen (bictegravir 50mg + tenofovir alafenamide 25 mg + emtricitabine 200 mg fixed dose combination) on the day of diagnosis. Those patients beginning immediate ART in the ED who are willing to have additional laboratory specimens drawn in the ED and become part of a cohort to receive ART and have ongoing biological specimens obtained and will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Suspected acute HIV infection
* agree to start immediate ART and to storage of laboratory specimens

Exclusion Criteria:

* Known chronic HIV infection
* severe renal or liver disease
* drug allergy/hypersensitivity
* prohibited medications
* pregnancy
* co-morbidity that the investigator feels would compromise safety, data interpretation, or achieving study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of immediate ART initiation | 1 day
  Proportion of participants that initiate immediate ART and collection of laboratory specimens at baseline for suspected acute HIV

SECONDARY OUTCOMES:
Impact on linkage and engagement in care | 48 weeks
  Proportion with immediate ART for individuals with suspected acute HIV infection with linkage and 48 week engagement in care
ART effects on cell associated HIV DNA | 48 weeks
  Changes in cell associated HIV DNA (assays TBD based on best practices at the time of study completion)
ART effects leukocytes | 48 weeks
  Changes in proportion of activated lymphocytes activated monocytes
ART effects inflammation | 48 weeks
  Changes C-reactive protein levels
ART effects monocyte activation | 48 weeks
  Changes in soluble cd14 levels

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Jacobson, MD, Study Chair — University of Southern California
Locations (2):
- United States (2):
  - LA County-USC Medical Center Emergency Department, Los Angeles, California
  - Rand Schrader Health and Research Clinic, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No